CLINICAL TRIAL: NCT03085329
Title: A Study to Evaluate the Efficacy of Seattle-PAP for the Respiratory Support of Premature Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Charles Smith, Professor of Pediatrics, Principal Investigator, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Seattle-PAP 002
Record Dates: First submitted 2017-03-06; First posted 2017-03-21 (Actual); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Premature Birth
Keywords: bubble nasal continuous positive airway pressure; respiratory support
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: With written informed consent from the mother or parents, infants born at less than 30 weeks gestation and who are capable of breathing spontaneously within the first 72 hours postnatal, will be supported by bubble nasal continuous positive airway pressure (Bn-CPAP), randomized to the standard device from Fisher & Paykel or to Seattle-PAP.
Masking Description: The nature of this comparative study makes masking device assignment impractical. The objectivity of the outcome assessment will rely upon adherence to formally defined criteria for device support failure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Seattle-PAP (Experimental): bubble nasal cpap respiratory support with Seattle-PAP bubbler device, with all other aspects of care per usual care noninvasive respiratory support
  Interventions: Device: Seattle-PAP
- Conventional bubble nasal CPAP (Experimental): qualified and enrolled infants randomized to this arm will receive noninvasive respiratory support by bubble nasal CPAP, using the Fisher & Paykel bubbler, which is the standard of care at Nationwide Children's.
  Interventions: Device: Conventional bubble nasal CPAP

INTERVENTIONS:
Device: Seattle-PAP — Seattle-PAP is a modified bubble CPAP device that has been given 510(k) clearance by the US FDA (K131502, October 11, 2013) and is thus recognized as substantially equivalent to other approved devices on the market. Results of a recently completed study in infants indicate that Bn-CPAP is associated with lower effort to breathe by spontaneously breathing premature infants.
  Arms: Seattle-PAP
Device: Conventional bubble nasal CPAP — Infants enrolled in the study and randomized to this arm will be given respiratory support by bubble nasal CPAP using the Fisher & Paykel bubbler device, which is the standard of care at Nationwide Children's.
  Arms: Conventional bubble nasal CPAP

SUMMARY:
This study is designed to test the hypothesis that among infants born at less than 30 weeks, weighing less than 1500 g at delivery, and receiving initial respiratory support non-invasively or on invasive respiratory support and meeting extubation criteria in the first 72 h of life, fewer neonates managed on Seattle--PAP will require endotracheal intubation and conventional mechanical ventilation (CMV) than will neonates managed from birth on bubble nasal continuous positive airway pressure (Bn-CPAP) using the Fischer- & Paykel (FP) device. Neonates on nasal continuous positive airway pressure (CPAP) in the delivery room or who are stabilized on mechanical ventilation as their initial form of respiratory support and meet our criteria for extubation within 72 h of birth will be eligible for randomization and study.

The primary endpoint of this study is the cumulative incidence of respiratory failure requiring intubation that occurs in patients after randomization and before 36 weeks post menstrual age (PMA) or discharge, whichever comes first. Presently, the literature supports that this age group typically exhibits intubation rates of 50% or more, which is consistent with the data from the Nationwide Children's Hospital/Ohio State University (NCH/OSU) Neonatal Intensive Care Unit (NICU).

DETAILED DESCRIPTION:
Parents / Mothers with impending pre-term delivery at <30 weeks of gestation will be approached for informed consent to participate. If consent is given prior to delivery, upon delivery the neonate may be randomly assigned to either Fisher & Paykel CPAP (conventional approach) or Seattle--PAP (experimental approach).

First 72 hours of life: 1) Neonates able to breathe spontaneously on less than 40% oxygen after initial resuscitative efforts and would normally be placed on CPAP will be randomly assigned to one of the two treatment groups using sealed cards generated by a variable block randomization scheme. 2) Neonates requiring increased support after initial resuscitation (intubation, >40% oxygen by CPAP) will not initially be randomized. However, if within the first 72 hours of life, the infant meets NCH criteria for extubation, randomization to CPAP delivery method will be performed. 3) Neonates born at <30 weeks gestation who were intubated at birth and are unable to be weaned from ventilator support will be removed from the study.

72 Hours - 32 Weeks of Life: 1) Neonates from the first period (First 72 Hours of Life, above) who remain on CPAP will continue on randomly assigned CPAP methodology. 2) Neonates from the first period, who failed stabilization on CPAP and required intubation, but are able to be extubated to CPAP will be placed back on their assigned CPAP method. 3) Attempts will be made to wean back to assigned CPAP method any neonates who are >72 hours old and require intubation beyond this period for any reason. 4) If unable to wean back to CPAP prior to 32 weeks of age, these patients will be removed from the study.

CPAP Failure (Sub-Group 1): For the neonates initially assigned to CPAP in the delivery room (sub-group 1), respiratory failure secondary to hyaline membrane disease is recognized as a common occurrence. If a patient assigned to this group, regardless of CPAP methodology, requires a fraction of inspired oxygen (FiO2) greater than 0.40 on CPAP of 6 cm of water (H2O), or is deemed to require intubation for adequate oxygenation, this will be considered a failure of CPAP stabilization. These patients, however, may remain in the study if it becomes clinically feasible to return them back to their assigned CPAP method prior to 72 hours of life. If this is unable to be done, they will be removed from the study.

CPAP Failure (Sub-Group 2): Any neonate that requires FiO2 greater than 0.40 on CPAP of 6 cm H2O or intubation beyond the first 72 hours of life will also be considered CPAP failures. Like those assigned to sub-group 1, these patients may remain in the study if it becomes clinically feasible to return them back to their assigned CPAP method prior to 32 weeks of life. If this is unable to be done, they will be removed from the study.

All patients who are not removed from the study as outlined above or due to other unforeseen circumstances will be monitored to discharge for any change in ventilation and ventilation requirement status. Routine care, including clinical exams and procedures (echocardiography, ultrasound, eye exams, x--rays) that would be considered standard of care for these patients will be performed at the medical discretion of the assigned care providers. No changes other than the type of CPAP device used (if applicable) will be necessary to routine practice.

Transfers to NCH: [From Outside Hospital] - Neonates born at an outside institution who meet the inclusion criteria (<30 weeks GA, able to spontaneously breathe by 72 hours of life or were initially placed on CPAP and failed, <32 weeks of age) and whose parents can be reached to obtain consent will be considered for inclusion in this research study. [Transfers from Ohio State University (OSU) Hospital] - It is recognized that many neonates born at OSU will require transport to NCH for further medical care. Having fulfilled inclusion criteria at OSU, transport to NCH will not result in removal from the study.

Cardiopulmonary Monitoring: All neonates are monitored in the NICU using pulse oximetry as part of normal practice. Many potential subjects in this study are also monitored through blood tests and arterial catheters, the latter of which are normally not intended for long term use.

Pressure Monitoring: A stand-alone Data Acquisition and Recording Instrument (DARCI) that measures pressure (i.e., positive airway pressure [PAW]) will be attached to the ventilation circuit. The DARCI unit is equipped with a standard International Organization for Standardization (ISO)19054 pole mount fitting attached on the back. A medical grade plug-in transformer provides electrical power (120 volts alternating current (AC) to 5 volts direct current (DC)). An internal battery and on-board non-volatile memory provide continuous data processing and storage in the event of power interruption or loss. A start button with a green light emitting diode (LED) and a stop button with a red LED provide the operational interface to the user during setup and changes in ventilation circuits. Initial programming and downloading of recorded pressure data will be accomplished using a laptop personal computer (PC) with interface application software installed.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent from parents, less than 30 weeks postmenstrual age at birth, within 72 h of postnatal age spontaneously breathing and able to sustain SaO2 of greater than 90% on less than or equal to FiO2 of 0.40 and 6 cm H2O pressure

Exclusion Criteria:

* Cardiopulmonary malformations (cardiac valve atresia, lung atresia)
* Congenital malformations (examples: anencephaly, omphalocele, Tetralogy of Fallot) Genetic anomalies (examples: Trisomy 21, Trisomy 18).

Max Age: 30 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 220 (Estimated)
Dates: Start 2017-02-10 (Actual); Primary Completion 2018-10-31 (Estimated); Study Completion 2019-02-09 (Estimated)

PRIMARY OUTCOMES:
Failure of noninvasive respiratory support | After randomization and before 36 weeks postmenstrual age (PMA) or discharge from the hospital, whichever comes first.
  The primary endpoint of this study is the cumulative incidence of respiratory failure requiring intubation. The principal criteria for failure of support are the requirement of an FiO2 greater than 0.40 and CPAP of greater than 6 cm H2O to maintain SaO2 of at least 90%. Support failure also can be declared by the responsible clinician based on best clinical judgment, but any declarations not based on the stated criteria will require written explanations.

SECONDARY OUTCOMES:
pneumothorax | After randomization and before 36 weeks postmenstrual age (PMA) or discharge from the hospital, whichever comes first.
  by diagnosis of clinical care team
nasal trauma | After randomization and before 36 weeks postmenstrual age (PMA) or discharge from the hospital, whichever comes first.
  by diagnosis of clinical care team
supplemental oxygen requirement | After randomization and before 36 weeks postmenstrual age (PMA) or discharge from the hospital, whichever comes first.
  if an infant fails for one hour or more fails to sustain an oxygen saturation (SaO2) of at least 90 percent, with FiO2 of 0.40 or less and 6 cm of water pressure (cmH2O) or less CPAP pressure.
ventilation-associated sepsis | After randomization and before 36 weeks postmenstrual age (PMA) or discharge from the hospital, whichever comes first.
  by diagnosis of clinical care team
death of infant | After randomization and before 36 weeks postmenstrual age (PMA) or discharge from the hospital, whichever comes first.
  infant declared dead by responsible clinical care personnel
Central nervous system (CNS) injury | After randomization and before 36 weeks postmenstrual age (PMA) or discharge from the hospital, whichever comes first.
  intraventricular hemorrhage and/or periventricular leukomalacia
gastrointestinal complications | After randomization and before 36 weeks postmenstrual age (PMA) or discharge from the hospital, whichever comes first.
  necrotizing enterocolitis and/or spontaneous intestinal perforation
retinopathy of prematurity | After randomization and before 36 weeks postmenstrual age (PMA) or discharge from the hospital, whichever comes first.
  by diagnosis of clinical care team

CONTACTS AND LOCATIONS:
Overall Officials: Carl H Backes, Jr., MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
The data will be available for download via Globus sharing services from the Seattle-PAP shared endpoint.

REFERENCES:
- [Background] Diblasi RM, Zignego JC, Tang DM, Hildebrandt J, Smith CV, Hansen TN, Richardson CP. Noninvasive respiratory support of juvenile rabbits by high-amplitude bubble continuous positive airway pressure. Pediatr Res. 2010 Jun;67(6):624-9. doi: 10.1203/PDR.0b013e3181dcd580. PMID 20308940
- [Result] Welty SE. Continuous Positive Airway Pressure Strategies with Bubble Nasal Continuous Positive Airway Pressure: Not All Bubbling Is the Same: The Seattle Positive Airway Pressure System. Clin Perinatol. 2016 Dec;43(4):661-671. doi: 10.1016/j.clp.2016.07.004. PMID 27837751
- [Result] Diblasi RM, Zignego JC, Smith CV, Hansen TN, Richardson CP. Effective gas exchange in paralyzed juvenile rabbits using simple, inexpensive respiratory support devices. Pediatr Res. 2010 Dec;68(6):526-30. doi: 10.1203/PDR.0b013e3181f985f0. PMID 20814347
- [Result] Kirpalani H, Millar D, Lemyre B, Yoder BA, Chiu A, Roberts RS; NIPPV Study Group. A trial comparing noninvasive ventilation strategies in preterm infants. N Engl J Med. 2013 Aug 15;369(7):611-20. doi: 10.1056/NEJMoa1214533. PMID 23944299
- [Derived] Backes CH, Notestine JL, Lamp JM, Balough JC, Notestine AM, Alfred CM, Kern JM, Stenger MR, Rivera BK, Moallem M, Miller RR, Naik A, Cooper JN, Howard CR, Welty SE, Hillman NH, Zupancic JAF, Stanberry LI, Hansen TN, Smith CV. Evaluating the efficacy of Seattle-PAP for the respiratory support of premature neonates: study protocol for a randomized controlled trial. Trials. 2019 Jan 18;20(1):63. doi: 10.1186/s13063-018-3166-6. PMID 30658678